CLINICAL TRIAL: NCT05237232
Title: Cerebral Hemodynamic Impact in Children Depending on the Technique of Carotid Artery Decanulation Technique After Extracorporeal Membrane Oxygenation: Modeling of Intra-cerebral Vascular Flows
Brief Title: Modeling of Intracerebral Vascularization After Extracorporeal Membrane Oxygenation in Children
Acronym: MoVa-ECMO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211306; 2021-A01935-36 (Other: IDRCB number)
Record Dates: First submitted 2022-01-28; First posted 2022-02-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Extra Corporeal Membrane Oxygenation; Decanulated Alive
Keywords: Extra corporeal membrane oxygenation; Pediatric patients; Arterial circulation; Techniques of carotid decanulation; Circle of Willis; Magnetic Resonance Angiography
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Newborns, infants and children hospitalized in pediatric intensive care unit (PICU) at Trousseau Hospital, having been treated with jugulocarotid ECMO and weaned alive off ECMO.
  Interventions: Other: Modeling cerebral vascularization
- Controls: Newborns treated for hypoxic-ischemic encephalopathy in the PICU of Trousseau Hospital.
  Interventions: Other: Magnetic Resonance Angiography (MRA) additional acquisition time; Other: Modeling cerebral vascularization

INTERVENTIONS:
Other: Magnetic Resonance Angiography (MRA) additional acquisition time — Additional acquisition time, time of flight, during brain MRA of the care allowing to obtain the same quality of vascular anatomical visualization as the brain MRA with gadolinium contrast medium injection performed for the care of the patients treated with jugulocarotid ECMO.
  Groups: Controls
Other: Modeling cerebral vascularization — The modeling of cerebral vascularization from CRIMSON software (CaRdiovascular Integrated Modeling & Simulation) requires several inputs:
  * The MRA images
  * The cardiac function curve
  * The cerebral blood flow
  * Measurement of systolic, diastolic and mean arterial blood pressure

SUMMARY:
Extra corporeal membrane oxygenation (ECMO) is a transient supplementation technique that alleviates hemodynamic and ventilatory failure. Its implementation requires carotid arterial and jugular venous cannulation in newborns or children weighing less than 20 kg. The impact of ECMO on arterial circulation was studied by Doppler ultrasound and shows a redistribution of flows within the circle of Willis.

This study aims to model cerebral flow in children who have been cared from jugulocarotid ECMO and compare cerebral hemodynamics according to the technique of reconstruction of the common carotid artery after decanulation (reconstruction or ligation).

DETAILED DESCRIPTION:
Extra corporeal membrane oxygenation (ECMO) is a transient supplementation technique that alleviates hemodynamic and ventilatory failure. Its implementation requires carotid arterial and jugular venous cannulation in newborns or children weighing less than 20 kg. The impact of ECMO on arterial circulation was studied by Doppler ultrasound and shows a redistribution of flows within the circle of Willis.

When ECMO is stopped, carotid decanulation is done either by ligation or by reconstruction, depending on the practices of the surgical team and the peroperative findings. The reconstruction allows a restoration of blood flow to the internal carotid artery and the middle cerebral artery with a disappearance of compensation by the circle of Willis.

Vascular flow modeling is a computational method derived from imaging for the hemodynamic study of fluids, including pressures and flow rates at different points in a vessel. Data from the literature on the modeling of cerebral vascularization in newborns are scarce.

This study aims to model cerebral flow in children who have been cared from jugulocarotid ECMO and compare cerebral hemodynamics according to the technique of reconstruction of the common carotid artery after decanulation (reconstruction or ligation).

ELIGIBILITY:
Inclusion Criteria:

For everyone :

1. Information and non-opposition of holders of parental authority
2. Newborn, infant and child <20kg
3. Hospitalization in pediatric and neonatal intensive care unit (PICU) of Trousseau Hospital
4. Performing a Magnetic Resonance Angiography (MRA) as part of the treatment

   For patients treated with ECMO: study population
5. Hemodynamic or respiratory failure
6. Requiring the use of extracorporeal circulation with jugulo-carotid cannulation
7. Weaned alive off Extra corporeal membrane oxygenation (ECMO)

   For patients with hypoxic-ischemic encephalopathy: control population
8. hypoxic-ischemic encephalopathy diagnosed at birth

Exclusion Criteria:

1. Contraindication to MRA
2. Opposition of holders of parental authority

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns, infants and children having been treated with jugulocarotid ECMO and weaned alive off ECMO and newborns treated for hypoxic-ischemic encephalopathy, hospitalized in pediatric intensive care unit (PICU) at Trousseau Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Intracerebral arterial flows of patients treated with ECMO | 1 month
  Comparison of intracerebral arterial flows according to the technique of reconstruction of the common carotid artery (reconstruction or ligation) after decanulation from data of MRA performed in weaned living patients off ECMO using computational fluid dynamic.

SECONDARY OUTCOMES:
Modeling of the flow of internal carotid arteries in their extra-cranial portion in children after ECMO | 1 month
  Brain Magnetic Resonance Angiography (MRA)
Cerebral vascularization of patients treated for hypoxic-ischemic encephalopathy | 1 month
  Additional acquisition time, time of flight, during brain Magnetic Resonance Angiography. (MRA) of the care.
  Modeling of the normal cerebral vascularization in children and infants / newborns.
Intracerebral arterial flows of patients treated for hypoxic-ischemic encephalopathy | 1 month
  Comparison of intracerebral arterial flows between patients treated with ECMO and those treated for anoxo-ischemia from data of MRA and by using computational fluid dynamic.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Irtan, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Garance Martin, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No